CLINICAL TRIAL: NCT00850252
Title: Use of a Completely Autologous and Completely Biological Tissue Engineered Blood Vessel Lifeline as an Arteriovenous Fistula in Hemodialysis Patients - Safety and Efficacy Study.
Brief Title: Use of a Lifeline Graft in the A-V Shunt Model
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cytograft Tissue Engineering (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cytograft A-V; R44HL064462-06 (NIH)
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: ESRD; Hemodialysis
Keywords: Lifeline; Tissue engineered blood vessel; A-V shunt
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Blood Vessel Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifeline blood vessel (Experimental)
  Interventions: Device: Lifeline

INTERVENTIONS:
Device: Lifeline — Surgical arteriovenous fistula formation with the use of Lifeline blood vessel
  Other Names: Tissue engineered blood vessel

SUMMARY:
This study will assess the safety and efficacy of a completely autologous and completely biological tissue engineered blood vessel (TEBV) called Lifeline™ used as an arteriovenous fistula for dialysis access.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an informed consent
* Patients ≥ 21 years old
* Patients not candidates for a Brescia-Cimino A-V fistula (own vessels)
* Have an AV shunt or fistula that will likely fail within 12 months because of:

  * Signs of clinical dysfunction: increment of venous pressure, limited site of puncture, stenosis, aneurysm dilatations that cannot be surgically repaired or by other media, or
  * Previous angioplasty, or
  * Previous thrombolysis
* Fall into category of ASA grade 2 or below (or UK equivalent)
* Are willing and able to comply with 2, 4, 6, 8, 10, 12, 16, 20, 24, 36 and 52 week follow up and able to comply with biannual follow up thereafter.

Exclusion Criteria:

* A need for urgent surgery
* Penicillin allergy
* Patients with uncontrolled hypertension
* Morbid obesity (> 300 lbs)
* Active systemic infection
* Contraindication for anticoagulation
* Coagulopathy
* Acute renal failure
* Connective tissue diseases (i.e. Marfan's syndrome)
* Pregnant or nursing
* Life expectancy < 1 year
* Participation in another study involving an investigational device or new drug
* Other medical, social or psychological issues that, in the opinion of the principal investigator, preclude them from receiving the treatment and the procedures/evaluations of the post-operative follow up
* Inability or unwillingness to comply with the scheduled follow-up visit

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary purpose of this study will be to gain preliminary safety experience with Lifeline blood vessel as an arteriovenous fistula | minimum 3 months

SECONDARY OUTCOMES:
The secondary purpose of the study is to assess the efficacy of the Lifeline blood vessel used as hemodialysis access in ESRD patients | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Luis M de la Fuente, MD, Principal Investigator — IADT, Buenos Aires, Argentina; Lech Cierpka, MD PhD, Principal Investigator — Department of General, Vascular and Transplant Surgery, Katowice, Poland
Locations (2):
- Instituto Argentino de Diagnostico y Tratamiento, Buenos Aires, Argentina
- Department of General, Vascular and Transplant Surgery, Katowice, Poland